CLINICAL TRIAL: NCT00955435
Title: Proteomic Analysis of the Combined Hormonal Therapy and Radiation Therapy for Localized Prostate Cancer
Brief Title: Study of Blood and Urine Samples in Patients With Newly Diagnosed Localized Prostate Cancer Treated With Hormone Therapy and Radiation Therapy. ICORG 06-15
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: CTRIAL-IE (ICORG) 06-15; CTRIAL-IE (ICORG) 06-15; EU-20921
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Non-interventional — Patients receive induction hormones* (bicalutimide and releasing-hormone agonist) for approximately 4 months prior to starting radiotherapy per standard treatment. Patients then receive radiotherapy consisting of 74 Gy up to a maximum of 81 Gy to the prostate gland per standard treatment.
Genetic: Protein expression analysis
Genetic: Proteomic profiling
Other: Laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and urine from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This clinical trial is studying blood and urine samples in patients with newly diagnosed localized prostate cancer treated with hormone therapy and radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Detect changes in serum and urine proteomic profiles that predict outcome in patients with newly diagnosed localized prostate cancer treated with hormonal therapy and radiotherapy.
* Identify prognostic and biochemical markers of early disease progression in patients treated with this regimen.
* Identify unique protein expression and temporal alterations, in these profiles, that facilitate understanding of the factors predicting relapse or toxicity.
* Identify molecular signatures that allow identification of targets for therapeutic intervention.

OUTLINE: This is a multicenter study.

Patients receive induction hormones* (bicalutimide and releasing-hormone agonist) for approximately 4 months prior to starting radiotherapy (per standard treatment). Patients then receive radiotherapy consisting of 74 Gy up to a maximum of 81 Gy to the prostate gland per standard treatment.NOTE: * Patients receiving short-term hormonal treatment for 4-8 months are eligible to participate in the trial.

Blood and urine samples are collected at baseline, and periodically during and after induction therapy for proteomic analysis.

After completion of study therapy, patients are followed up periodically for 5 years and yearly thereafter for the duration of the trial.

ELIGIBILITY:
Inclusion criteria:

1. Age 18 years or over.
2. Histologically confirmed invasive adenocarcinoma of the prostate (by TURP or TRUS).
3. Localised prostate cancer with a Gleason score 7
4. Short term hormonal treatment 4-8 months
5. Performance status of KPS ≥ 60 / WHO 0-2
6. Absence of distant metastases

Exclusion criteria:

1. The patient has previously received treatment for prostate cancer other than TURP/ TRUS
2. The patient has had a bilateral orchidectomy
3. The patient has previously received hormonal treatment for prostate cancer
4. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the trial. In the opinion of the investigator, any evidence of severe or uncontrolled systematic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease
5. The patient has or had other co-existing malignancies within the past 5 years other than non- melanoma skin cancer
6. Treatment with non-approved or investigational drug within 30 days before day one of the trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with localised prostate cancer who will receive radiation therapy plus hormonal therapy, for 4 - 8 months, are eligible for the trial. Patients will be eligible to participate in the trial provided they have not received prior therapy for their prostate cancer. It is planned that 60 patients will participate in the research study. All patients will receive approx 4 months of induction hormone therapy (LHRH agonist and Bicalutamide) prior to starting radiotherapy treatment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2006-02 (Actual)

PRIMARY OUTCOMES:
Changes in serum and urine proteomic profiles | Ongoing until patient progression
Prognostic and biochemical markers of early disease progression | Ongoing until patient progression
Protein expression and temporal alterations | Ongoing until patient progression
Molecular targets | Ongoing until patient progression

CONTACTS AND LOCATIONS:
Overall Officials: John Gerard Armstrong, MD, MB, MRCPI, Principal Investigator — Saint Luke's Hospital
Locations (2):
- Ireland (2):
  - Beacon Hospital, Dublin
  - Saint Luke's Radiation Oncology Network, Dublin